CLINICAL TRIAL: NCT06142175
Title: A Real World Study of Treatment of Relmacabtagene Autoleucel in Relapsed or Refractory Large B-Cell Lymphoma
Brief Title: Relmacabtagene Autoleucel in Patients With LBCL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JWCAR029-008
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-11

CONDITIONS: Large B-cell Lymphoma
Keywords: Relmacabtagene Autoleucel; Chimeric antigen receptor T cells
MeSH Terms: interventions — relmacabtagene autoleucel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relmacabtagene Autoleucel: Relmacabtagene Autoleucel administered as a single IV infusion at a target dose of 1 x 10^8 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells on Day1.
  Interventions: Biological: Relmacabtagene Autoleucel

INTERVENTIONS:
Biological: Relmacabtagene Autoleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells
  Other Names: JWCAR029

SUMMARY:
To evaluate the efficacy and safety of Relmacabtagene autoleucel for the treatment of adult patients with relapsed or refractory (r/r) large B-cell lymphoma (LBCL) in real-world

DETAILED DESCRIPTION:
This is a post-marketing, multicenter, observational real-world study, including prospective and retrospective studies. The purpose of this study is to collect efficacy and safety data over a 6-month period following treatment of adult patients with r/r LBCL with Relmacabtagene autoleucel. The treating physicians in the study will determine the most appropriate diagnostic and therapeutic regimen for their patients based on clinical practice.There will be no therapeutic intervention as a result of this study. There will be no subgroups of any kind in this study, and subgroup analyses will be performed based on the actual data collected during the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with established r/r LBCL;
2. Patients already treated with commercially available Relmacabtagene Autoleucel

Exclusion Criteria:

No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: r/r LBCL
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  Percentage of participants with CR or PR

SECONDARY OUTCOMES:
CRR | 6 months
  Complete response rate
DOR | 6 months
  Duration of response
Progression-Free Survival (PFS) | 6 months
  PFS is defined as the time from the Relmacabtagene Autoleucel infusion date to the date of disease progression per Lugano classification or death from any cause.
Overall Survival (OS) | 6 months
  OS is defined as the time from Relmacabtagene Autoleucel infusion to the date of death from any cause.
Adverse events (AEs) | 6 months
  Types, frequency, and severity of adverse events and laboratory anomalies Physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, PhD, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Huiqiang Huang, PhD, Principal Investigator — Sun Yat-sen University; Liang Huang, PhD, Principal Investigator — Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, China; Ping Li, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine; Heng Mei, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Hongmei Jing, Principal Investigator — Peking University Third Hospital; Wenbin Qian, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Depei Wu, Principal Investigator — The First Affiliated Hospital of Soochow University; Ying Lu, Principal Investigator — Ningbo University People's Hospital; Huilai Zhang, Principal Investigator — Tianjin Cancer Hospital; Qingyuan Zhang, Principal Investigator — Harbin Medical University Tumor Hospital; Dehui Zou, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences; Yao Liu, Principal Investigator — Chongqing University Cancer Hospital; Jianqiu Wu, Principal Investigator — Jiangsu Provincial Tumor Hospital; Yajun Li, Principal Investigator — Hunan Cancer Hospital; Ru Feng, Principal Investigator — Southern Medical University, China; Yuhua Li, Principal Investigator — Nanfang Hospital, Southern Medical University; Zhifeng Li, Principal Investigator — The First Hospital of Xiamen University
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No